CLINICAL TRIAL: NCT03454386
Title: Use of the Stress Management and Resilience Training (SMART) Program in the Management of Irritable Bowel Syndrome: A Pilot Study
Brief Title: SMART Program in Irritable Bowel Syndrome (IBS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Lin Chang, MD, Co-Director, G. Oppenheimer Center for Neurobiology of Stress and Resilience, Vatche and Tamar Manoukian Division of Digestive Diseases, University of California, Los Angeles
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB#18-000235
Record Dates: First submitted 2018-02-26; First posted 2018-03-05 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome (IBS); Stress; Resilience; Stress Management and Resilience Training Program (SMART)
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Active Comparator): Stress Management and Resilience Training Program
  This group will be initially enrolled in the program.
  Interventions: Behavioral: Stress Management and Resilience Training Program
- Control (Other): Self-Management Stress Reduction Program
  This group will be placed in a self-management stress reduction program. During this time these participants will be given a popular stress reduction book to read over 12 weeks. They will complete questionnaires at weeks 4 and 12. After the 12 weeks, this group will be enrolled in the online SMART program and complete assessments at week 24 (upon completion of the program.
  Interventions: Behavioral: Self-Management Stress Reduction Program

INTERVENTIONS:
Behavioral: Stress Management and Resilience Training Program — This program targets attention and interpretation of events, people and the world through the skills of gratitude, compassion, acceptance, forgiveness and understanding of a higher meaning. The program involves two phases. The 4 week "training phase" begins with a group session that discusses the practices that can be used to enhance awareness and engagement through the principles listed above. Participants will receive twice weekly emails with videos that described a different practice for participants to use in their daily lives. The second phase is the "sustain phase" that is 8 weeks in duration. Participants are expected to continue using the daily practices learned during the training phase. Weekly emails will be sent with ways to incorporate these practices into their daily lives.
  Other Names: SMART Program
  Arms: Active Treatment
Behavioral: Self-Management Stress Reduction Program — Program participants will be given a popular stress reduction book to read over a 12 week period. Upon completion of this, they will be enrolled in the online SMART program for 12 weeks.
  Arms: Control

SUMMARY:
This is a pilot study to determine the efficacy of the Stress Management and Resilience Training (SMART) program in improving gastrointestinal and psychological symptoms, health-related quality of life, and satisfaction of care in patients with irritable bowel syndrome (IBS). Half of the participants will be enrolled in the SMART program initially. The other half will be placed in a self-management stress reduction program where they will read a popular stress reduction book over 12 weeks. Then they will have access to participate in the online SMART program.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a functional gastrointestinal disorder characterized by abdominal pain related to defecation and associated with changes in stool frequency and/or form. IBS is a stress sensitive disorder and its severity has been shown to be moderated by both acute and chronic stress. Furthermore, resilience, which is defined as the ability to positively adapt and thrive in the presence of stressors and adversity, has been shown to be lower in those with IBS and associated with more severe symptoms. Therapies aimed at stress reduction in IBS have been found to be effective in the management of IBS. To our knowledge, there are no reports in the literature of a therapy to target resilience in the IBS patient population.

The Stress Management and Resilience Training (SMART) program was developed by Dr. A. Sood at the Mayo clinic to reduce stress, decrease symptoms related to stress and enhance resiliency. This is accomplished by targeting human attention and interpretation of events, people and the world. Furthermore, methods to strengthen the skills of gratitude, compassion, acceptance, forgiveness and understanding of a higher meaning are taught. Previous studies have demonstrated that this program can improve stress, anxiety, resilience and quality of life of participants.

ELIGIBILITY:
Inclusion Criteria:

* Those with a diagnosis of IBS based on the Rome IV diagnostic criteria (recurrent abdominal pain at least once per week in the last 3 months associated with 2 of the following: related to defecation, associated with a change in stool frequency, associated with a change in stool form. Symptoms must have started 6 months prior to presentation)
* Between the ages of 18 and 70
* English speaking
* Are able to provide written, informed consent
* At least moderate IBS symptoms (based on an IBS symptom severity scale score [IBS-SSS] of 175 or higher)
* At least moderate levels of perceived stress (based on a perceived stress score of 14 or higher
* If receiving pharmacologic therapy for IBS, they must be on a stable dose for 30 days prior to enrollment

Exclusion Criteria:

* History of gastrointestinal disease including celiac disease, cirrhosis, gastrointestinal malignancy, inflammatory bowel disease
* History of gastrointestinal surgery (except appendectomy and cholecystectomy or gallbladder removal >6 months ago)
* Poorly controlled psychiatric disease such as severe depression (with or without suicidal ideation), severe anxiety, schizophrenia, dementia
* Currently receiving, or have received in the last 6 months, other stress reduction therapies such as mindfulness based stress reduction, meditation
* Excessive alcohol intake (up to 1 drink per day for females and 2 drinks per day for males)
* Illicit substance use
* High dose opiate use
* Pregnancy
* Non-English speaking
* Inability to provide written informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Change in perceived stress score from baseline | Week 12 (end of the SMART program)
  Validated questionnaire with 10 questions regarding respondents stress levels

SECONDARY OUTCOMES:
Change in perceived stress score from baseline | Week 4
  Validated questionnaire with 10 questions regarding respondents stress levels
IBS symptom severity responder rate | Week 4, week 12
  IBS symptom severity will be measured using the validated IBS symptom severity score. A participant will be consider a responder if they have a 50 point reduction in their baseline score.
IBS related quality of life responder rate | Week 4, week 12
  IBS related quality of life will be measure using a validated questionnaire. A participant is considered a responder if there is a 14 point improvement in their baseline score
Change from baseline in resilience scores as measured by the Brief Resilience scale | Week 4, week 12
  The Brief Resilience scale is a 6 question validated questionnaire
Change from baseline in resilience score as measured by the Connor-Davidson Resilience Scale | Week 4, week 12
  The Connor-Davidson Resilience Scale is a 25 question validated questionnaire
Change from baseline in adaptive resilience score | Week 4, week 12
  A validated questionnaire to measure adaptive resilience will be used
Change in gratitude scores from baseline | Week 4, week 12
  Gratitude will be measured using a validated questionnaire.
Change in mindfulness scores from baseline | Week 4, week 12
  Mindfulness will be measured using the validated five factor mindfulness questionnaire
Change in patient satisfaction from baseline | Week 4, week 12
  The measurement of patient satisfaction will be adapted from the patient global satisfaction scale from the Hospital Consumer Assessment of Healthcare Providers and Systems.
Change in anxiety symptoms from baseline | Week 4, week 12
  Anxiety symptoms will be measured using the validated hospital anxiety and depression questionnaire
Change in gastrointestinal symptom related anxiety from baseline | Week 4, week 12
  Gastrointestinal symptom related anxiety will be measured using the validated visceral sensitivity index
Change in somatic symptom severity from baseline | Week 4, week 12
  Somatic symptom severity will be measured using the validated patient health questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lin Chang, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States